CLINICAL TRIAL: NCT03328429
Title: Comparison of Intraoperative and Postoperative Outcomes of Bartholin Gland Marsupialisation Versus Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Attending physician,ObGyn, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/220
Record Dates: First submitted 2017-10-22; First posted 2017-11-01 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Bartholin Abscess
Keywords: bartholin; marsupialisation; abscess
MeSH Terms: conditions — Abscess

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marsupialization (Other): Bartholin gland marsupialization will be done to all patients with Bartholin abscess.
  Interventions: Other: Marsupialization
- Excision (Other): Bartholin gland excision will be done to all patients with Bartholin abscess.
  Interventions: Other: Excision

INTERVENTIONS:
Other: Excision — Bartholin gland will be excised
  Arms: Excision
Other: Marsupialization — Bartholin gland will be marsupialised
  Arms: Marsupialization

SUMMARY:
To compare intraoperative and postoperative outcomes of Bartholin marsupialisation versus excision

DETAILED DESCRIPTION:
Bartholin cysts and abscess are commonly seen. Different surgical procedures are done for therapy. Our aim is to compare intraoperative results and postoperative healing of patients undergoing marsupialisation versus excision.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40, Bartholin cyst/abscess

Exclusion Criteria:

* patients with systemical diseases, patients with recurrent Bartholin abscess

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients with Bartholin cyst/abscess
Enrollment: 154 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
postoperative | 3 months
  Patients will be followed up for three months. 3 months after the surgery, all patients will be asked to complete the Female Sexual Function Index (FSFI) questionnaire alone in a hospital room. The FSFI includes a total of 19-item validated questionnaire which was used for the evaluation of sexual desire, arousal, lubrication, orgasm, satisfaction, and pain during sexual intercourse. Scores range from 2 to 36, higher scores indicate better sexual function. Sexual dysfunction is described as having a total FSFI score of 26.55 or less.

SECONDARY OUTCOMES:
operation time | during procedure
  operation time during the procedure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aslan Çein, Principal Investigator — KSSTRH
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ozdegirmenci O, Kayikcioglu F, Haberal A. Prospective Randomized Study of Marsupialization versus Silver Nitrate Application in the Management of Bartholin Gland Cysts and Abscesses. J Minim Invasive Gynecol. 2009 Mar-Apr;16(2):149-52. doi: 10.1016/j.jmig.2008.10.006. PMID 19598336